CLINICAL TRIAL: NCT03845699
Title: Development of an Algorithm That Predicts Hypoventilation Due to an Opioid Overdose
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RTM Vital Signs, LLC (Industry)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 20183438,18C.7
Record Dates: First submitted 2019-02-16; First posted 2019-02-19 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Drug Overdose; Opioid-Related Disorders
Keywords: Opioid Overdose; Diagnostic Algorithm; Wearable Trachea Sound Sensor; Respiratory Depression; Hypoventilation
MeSH Terms: conditions — Drug Overdose; Opioid-Related Disorders; Opiate Overdose; Respiratory Insufficiency; Hypoventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Diagnostic algorithms that detects/predicts hypoventilation — Produce mild and moderate respiratory depression (hypoventilation) using a controlled intravenous infusion of fentanyl while measuring/recording respiratory rate, tidal volume, body activity, and body position.
  Other Names: Infusion of fentanyl to induce hypoventilation

SUMMARY:
RTM Vital Signs, LLC is developing a miniature wearable tracheal sound sensor that communicates with a cell phone containing a machine-learning diagnostic algorithm designed to detect and predict the onset of mild, moderate, and severe hypoventilation (respiratory depression) due to an opioid overdose. The purpose of this clinical trial is to develop/validate diagnostic algorithms capable of detecting/predicting the onset of hypoventilation induced by a controlled intravenous infusion of fentanyl. The wearable sensor and algorithms will provide a series of alerts and alarms to the person, caregiver, and/or emergency personnel.

DETAILED DESCRIPTION:
More than 64,000 Americans died from a drug overdose in 2016 and drug overdose is now the most common cause of death for people under 50 years old in the United States. The purpose of this study is to design a wearable tracheal sound sensor and develop an experimental computer program (diagnostic algorithm) that can accurately detect and predict the onset of mild, moderate, and severe hypoventilation (slow and shallow breathing) due to an opioid (fentanyl) overdose

Opioid pain medications routinely cause a person's breathing to become slower and shallower, leading to an increased amount of carbon dioxide and decreased amount of oxygen in the bloodstream. Microphone trachea sound sensors will be used to measure and record sounds produced by air movement in and out of a person's trachea (windpipe) during inhalation and exhalation. Blood will be frequently sampled from a catheter placed within a wrist artery to measure the concentration of carbon dioxide and oxygen. An intravenous infusion of fentanyl will be used to decrease the person's respiratory rate and depth of breathing over a 1 to 3 hour period. Other sensors will be used to accurately measure and record the person's respiratory rate, tidal volume, hemoglobin oxygen saturation, electrocardiogram, blood pressure, temperature, body activity level, and body position. Each sensor's output signal will be processed and filtered to enhance the signal-to-noise ratio. The Trachea Sound Sensor and reference respiratory sensor information will be used to develop/validate risk-index algorithms that can recognize a significant change in an individual's "normal or baseline" pattern of respiratory rate, tidal volume, body activity, and body position. The hypoventilation monitoring system will not require previous knowledge of an individual's age, height, weight, model of the respiratory tract, or external calibration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women/men between 18 and 40 years of age.
2. Negative history of drug or alcohol abuse.
3. Negative history of cigarette smoking in previous 6 months.
4. Negative history of active cardiac, vascular, pulmonary, renal, hepatic, nervous, metabolic or immune disease.
5. BMI < 30

Exclusion Criteria:

1. Age < 18 years and > 40 years.
2. Pregnant or planning to become pregnant.
3. Positive history drug or alcohol abuse.
4. Positive drug screen for opioids, benzodiazepines, hypnotics.
5. Positive Drug Abuse Screening Test result (score of 6 or greater).
6. BMI > 30
7. History of sleep apnea.
8. History of cigarette smoking in previous 6 months.
9. History of difficult airway during anesthesia management.
10. History of allergy or skin sensitivity to tape, silicone, fentanyl, chlorhexidine.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy males/females of all ethnic backgrounds, 18 to 40 years of age
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2020-05-14 (Estimated); Study Completion 2020-05-14 (Estimated)

PRIMARY OUTCOMES:
Percent Sensitivity and Specificity of Detecting/Predicting the Onset of Mild Hypoventilation due to an Opioid Overdose | 1 to 3 hours
  The investigators will evaluate the risk-index algorithm's ability to detect/predict at which point during the standardized fentanyl infusion protocol does mild hypoventilation actually occur. Calculate the percent sensitivity and specificity of detecting/predicting the onset of mild hypoventilation (PaCO2- 45 to 50 mm Hg) due to a fentanyl overdose.
Percent Sensitivity and Specificity of Detecting/Predicting the Onset of Moderate Hypoventilation due to an Opioid Overdose | 1 to 3 hours
  The investigators will evaluate the risk-index algorithm's ability to detect/predict at which point during the standardized fentanyl infusion protocol does moderate hypoventilation actually occur. Calculate the percent sensitivity and specificity of detecting/predicting the onset of mild hypoventilation (PaCO2- 51 to 60 mm Hg) due to a fentanyl overdose.
Percent Sensitivity and Specificity of Detecting/Predicting the Onset of Severe Hypoventilation due to an Opioid Overdose | 1 to 3 hours
  The investigators will evaluate the risk-index algorithm's ability to detect/predict at which point during the standardized fentanyl infusion protocol does severe hypoventilation actually occur. Calculate the percent sensitivity and specificity of detecting/predicting the onset of severe hypoventilation (PaCO2 > 60 mm Hg) due to a fentanyl overdose.

SECONDARY OUTCOMES:
Absolute Difference Between Trachea Sound Sensor's Measurements and Reference Sensor Measurements | 1 to 3 hours
  Correlation between the trachea sound sensor's measurements and the reference sensor measurements of respiratory rate, tidal volume, activity level, and body position during an intravenous infusion of fentanyl (Bland-Altman plot of absolute difference).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen McNulty, DO, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mildh LH, Scheinin H, Kirvela OA. The concentration-effect relationship of the respiratory depressant effects of alfentanil and fentanyl. Anesth Analg. 2001 Oct;93(4):939-46. doi: 10.1097/00000539-200110000-00028. PMID 11574361
- [Background] Boyer EW. Management of opioid analgesic overdose. N Engl J Med. 2012 Jul 12;367(2):146-55. doi: 10.1056/NEJMra1202561. No abstract available. PMID 22784117
- [Background] Volkow ND, Collins FS. The Role of Science in Addressing the Opioid Crisis. N Engl J Med. 2017 Jul 27;377(4):391-394. doi: 10.1056/NEJMsr1706626. Epub 2017 May 31. No abstract available. PMID 28564549
- [Background] Yadollahi A, Moussavi ZM. Acoustical respiratory flow. A review of reliable methods for measuring air flow. IEEE Eng Med Biol Mag. 2007 Jan-Feb;26(1):56-61. doi: 10.1109/memb.2007.289122. No abstract available. PMID 17278773
- [Background] Chen G, de la Cruz I, Rodriguez-Villegas E. Automatic lung tidal volumes estimation from tracheal sounds. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:1497-500. doi: 10.1109/EMBC.2014.6943885. PMID 25570253
- [Background] Ramsay MA, Usman M, Lagow E, Mendoza M, Untalan E, De Vol E. The accuracy, precision and reliability of measuring ventilatory rate and detecting ventilatory pause by rainbow acoustic monitoring and capnometry. Anesth Analg. 2013 Jul;117(1):69-75. doi: 10.1213/ANE.0b013e318290c798. Epub 2013 Apr 30. PMID 23632055
- [Background] Reyes BA, Reljin N, Chon KH. Tracheal sounds acquisition using smartphones. Sensors (Basel). 2014 Jul 30;14(8):13830-50. doi: 10.3390/s140813830. PMID 25196108
- [Background] Stuth EA, Stucke AG, Zuperku EJ. Effects of anesthetics, sedatives, and opioids on ventilatory control. Compr Physiol. 2012 Oct;2(4):2281-367. doi: 10.1002/cphy.c100061. PMID 23720250
- [Background] O'Croinin D, Ni Chonghaile M, Higgins B, Laffey JG. Bench-to-bedside review: Permissive hypercapnia. Crit Care. 2005 Feb;9(1):51-9. doi: 10.1186/cc2918. Epub 2004 Aug 5. PMID 15693984
- [Background] Vannucci RC, Towfighi J, Brucklacher RM, Vannucci SJ. Effect of extreme hypercapnia on hypoxic-ischemic brain damage in the immature rat. Pediatr Res. 2001 Jun;49(6):799-803. doi: 10.1203/00006450-200106000-00015. PMID 11385141
- [Background] Yu L, Ting CK, Hill BE, Orr JA, Brewer LM, Johnson KB, Egan TD, Westenskow DR. Using the entropy of tracheal sounds to detect apnea during sedation in healthy nonobese volunteers. Anesthesiology. 2013 Jun;118(6):1341-9. doi: 10.1097/ALN.0b013e318289bb30. PMID 23407106
- [Background] Penzel T, Sabil A. The use of tracheal sounds for the diagnosis of sleep apnoea. Breathe (Sheff). 2017 Jun;13(2):e37-e45. doi: 10.1183/20734735.008817. PMID 29184596
- [Background] Jin F, Goh DY, Louis IM. An Enhanced Respiratory Rate Montoring Method for Real Tracheal Sound Recordings. 17 European Signal Processing Conference. 2009:642- 645.
- [Background] Harper VP, Pasterkamp H, Kiyokawa H, Wodicka GR. Modeling and measurement of flow effects on tracheal sounds. IEEE Trans Biomed Eng. 2003 Jan;50(1):1-10. doi: 10.1109/TBME.2002.807327. PMID 12617519
- [Background] Bureev AS, Dikman EY, Zhdanov DS, Zemlyakov IY, Kutsov MS. Mathematic Model for Spectral Characteristics of Respiratory Sounds Registered in Trachea Region. Global Journal of Pure and Applied Mathematics. 2016;12(5):4569-4578.
- [Background] Kraman SS, Wodicka GR, Pressler GA, Pasterkamp H. Comparison of lung sound transducers using a bioacoustic transducer testing system. J Appl Physiol (1985). 2006 Aug;101(2):469-76. doi: 10.1152/japplphysiol.00273.2006. Epub 2006 Apr 20. PMID 16627681
- [Background] Lu BY. Unidirectional Microphone based Wireless Recorder for the Respiration Sound. J Bioengineer & Biomedical Sci. 2016;6(3).
- [Background] Perus O, Marsot A, Ramain E, Dahman M, Paci A, Raucoules-Aime M, Simon N. Performance of alfentanil target-controlled infusion in normal and morbidly obese female patients. Br J Anaesth. 2012 Oct;109(4):551-60. doi: 10.1093/bja/aes211. Epub 2012 Jun 24. PMID 22732112
- [Background] Shafer SL, Varvel JR, Aziz N, Scott JC. Pharmacokinetics of fentanyl administered by computer-controlled infusion pump. Anesthesiology. 1990 Dec;73(6):1091-102. doi: 10.1097/00000542-199012000-00005. PMID 2248388

DOCUMENTS (1):
  • Study Protocol (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT03845699/Prot_000.pdf